CLINICAL TRIAL: NCT04524520
Title: COVID19-OR (SARS-CoV-2):Observation, Risk & Recovery. An Observational Study Exploring Risk Assessment and Recovery From COVID-19 (SARS-CoV-2) Infection in Hospitalised Patients
Brief Title: COVID19-OR (SARS-CoV-2): Observation,Risk & Recovery
Status: Completed | Type: Observational
Sponsor: Western Sussex Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20/YH/0157
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Exploring Risk Assessment and Recovery From COVID-19 Infection in Hospitalised Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A novel coronavirus, designated corona virus disease 2019 (COVID-19) has resulted in a Pandemic at the time of writing (27th April) the reported number of confirmed cases exceeding 3 million and over 200000 associated deaths.

The burden on global critical care has been considerable. As of 24th April there have been 8752 UK critical care admissions with services under considerable strain, and a mortality rate over 50%. Survivors of critical illness will require significant input.

This study will perform mixed methods to provide rich data on risk stratification and recovery from critical illness. Recovery from a novel disease requires documenting and the study reports physical and psychological changes following hospital discharge in survivors. In addition qualitative interviews are being conducted with patients who have survived and been discharged from critical care along with their relatives and treating professionals, to better understand their needs during recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years admitted to ICU with SARS-CoV-2 and survived
2. Relatives or friends and professionals involved in the care of these patients.

Exclusion Criteria:

1. Patients <18 years;
2. Patients with a negative test for SARS-CoV-2 or patients not tested due to absence of symptoms;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to hospital with suspected/confirmed COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Physical | through study completion , an average of 1 year
  Chelsea critical care physical assessment tool
Physical | through study completion , an average of 1 year
  Incremental Shuttle Walk Test (ISWT)
Physical | through study completion , an average of 1 year
  1- minute Sit to Stand, Grip strength
Health Related Quality of life | at 3 months
  Short Form Survey on health related quality of life (SF-12). Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. Higher scores indicate better outcome.
Health Related Quality of life | at 1 year
  Short Form Survey on health related quality of life (SF-36). Scores can range from 0 to 100 and a higher score indicates better outcome.
Psychological | through study completion , an average of 1 year
  Depression Test Questionnaire (PHQ-9). Scores range from 1 to 27 and higher scores indicate worse outcome.
Psychological | through study completion , an average of 1 year
  Anxiety Test Questionnaire (GAD-7). Scores range from 0 to 21 and higher scores indicates worse outcome.
Psychological | through study completion , an average of 1 year
  Montreal Cognitive Assessment (MoCA). Scores range from 0 to 30 and higher scores indicate a better outcome.
Psychological | at 1 year
  Post-traumatic stress disorder (PTSD) Trauma Screening (TSQ). A screening tool with 10 items. If 6 items are endorsed then the outcome is 'positive' for PTSD.

SECONDARY OUTCOMES:
risk stratification | through study completion and average of 1 year
  escalation to critical care (Yes/No)
risk stratification | through study completion and average of 1 year
  mechanical ventilation (Yes/No)
risk stratification | through study completion and average of 1 year
  critical care stay hospital stay (number of days)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Luke Hodgson, Principal Investigator — Western Sussex Hospitals NHS Trust
Locations (1):
- Dr Luke Hodgson, Worthing, United Kingdom